CLINICAL TRIAL: NCT06217848
Title: The Effect of GLP-1 Agonist in Patients With Hypothalamic Obesity: Prospective, Pilot Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hee Kim, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2208-031-1348
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Panhypopituitarism; Craniopharyngioma; Hypothalamic Obesity
MeSH Terms: conditions — Combined Pituitary Hormone Deficiency; Craniopharyngioma; Sexual Infantilism | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients diagnosed with a hypothalamic tumor. (Experimental)
  Interventions: Drug: Saxenda

INTERVENTIONS:
Drug: Saxenda — Patients will receive subcutaneous injections of Saxenda 18 mg/3 mL Pen (liraglutide_obesity) starting at 0.6 mg qd. Increase by 0.6 mg qd at weekly intervals to 1.2 mg qd in week 2, 1.8 mg qd in week 3, 2.4 mg qd in week 4, 3.0 mg qd in week 5, and maintain for 8 weeks at a maximally tolerated dose within 3.0 mg starting in week 5. If the subject's response to treatment does not allow for escalation to the planned dose, subjects will inject an adaptive maximally tolerated dose within the planned dose at each cycle. Total duration of Saxenda treatment is 12 weeks.

SUMMARY:
GLP-1 analogs are used as agents in the existing treatment of obesity. However, there are lack of previous reports on the effectiveness and role of GLP-1 analogs in the development of obesity traits in patients with functionally impaired hypothalamus. With this preliminary study, the investigators would explore the role of GLP-1 analogues to identify eating behavioral pathology subtype differences in the therapeutic efficacy of GLP-1 analogues in hypothalamic obesity patients. This will allow us to identify the role of specific nuclei which could be the pathogenesis of hypothalamic obesity.

Our hypotheses: GLP-1 analogs will effectively induce weight loss in patients with hypothalamic obesity, and different subtypes of hypothalamic obesity will respond differently to GLP-1 analogs.

DETAILED DESCRIPTION:
Study Overview

* Collecting baseline clinical information, comorbidities, pituitary hormone status assessment, and treatment options, including supplemental therapies and surgery.
* Assessment of factors associated with obesity through physical measurements, questionnaires, and cognitive-behavioral tasks, and division of patients by eating behavior subtypes for further analysis.
* Collecting patients' meal records and meal times by self-reporting.
* Collecting data on patients' activity and sleep patterns through wearable devices.
* Patients will receive subcutaneous injections of Saxenda 18 mg/3 mL Pen (liraglutide_obesity) starting at 0.6 mg qd. Increase by 0.6 mg qd at weekly intervals to 1.2 mg qd in week 2, 1.8 mg qd in week 3, 2.4 mg qd in week 4, 3.0 mg qd in week 5, and maintain for 8 weeks at a maximally tolerated dose within 3.0 mg starting in week 5. If the subject's response to treatment does not allow for escalation to the planned dose, subjects will inject an adaptive maximally tolerated dose within the planned dose at each cycle. Total duration of Saxenda treatment is 12 weeks.

Eating behavior assessment questionnaires and cognitive behavioral tasks will be completed before the first dose, before the end of the dose escalation period, and after the final dose to explore treatment response.

Study Eligibility

- Patients aged 19 years and older who were diagnosed with a hypothalamic tumor and surgically treated at Seoul National University Hospital, and who met the inclusion and exclusion criteria after receiving a full explanation of the study and voluntary consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a hypothalamic tumor and treated surgically with confirmed hypothalamic damage
* 19 years of age or older
* Have a body mass index of at least 27 and less than 30 (27≤BMI<30) and one or more confirmed weight-related medical conditions, or a body mass index of 30 or greater (BMI≥30).
* Voluntarily agreed to participate in the study after receiving a full explanation of the study.

Exclusion Criteria:

* Unable to fully understand the instructions for participation in the study or unable to give voluntary consent.
* Presence or history of a medical condition or disease that, in the opinion of the investigator, would make it difficult for the patient to participate fully for the duration of the study or to interpret the results of the study
* Taking medications that may affect weight, except for hormone replacement therapy, in the last 6 months
* non-primary tumor patient
* Diagnosis of severe renal dysfunction, liver dysfunction, or thyroid disease among other underlying conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea